CLINICAL TRIAL: NCT00035464
Title: Efficacy and Safety of Azimilide in the Prophylactic Treatment of Patients
Brief Title: Efficacy and Safety of Azimilide in the Prophylactic Treatment of Patients With Atrial Fibrillation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Martin Phillips, MD, Procter & Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000037
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — azimilide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo
- 2 (Experimental): 125 mg azimilide tablets
  Interventions: Drug: Azimilide Dihydrochloride

INTERVENTIONS:
Drug: Azimilide Dihydrochloride — 125 mg azimilide tablets, twice a day for 6 months
  Arms: 2
Drug: Placebo — placebo tablets, twice a day for 6 months
  Arms: 1

SUMMARY:
Atrial fibrillation (an abnormal rhythm in the upper chamber of the heart) is a common supraventricular arrhythmia (a type of abnormal heart rhythm) for which antiarrhythmic therapy is often prescribed. The primary goals of therapy are to maintain sinus rhythm (normal heart rhythm) and to reduce the occurrence of episodes of atrial fibrillation. Azimilide may have an effect on increasing the time to first recurrence of symptomatic atrial fibrillation or atrial flutter and symptomatic paroxysmal supraventricular tachycardia (other types of abnormal heart rhythms).

This double-blind, placebo-controlled study is designed to evaluate the efficacy and safety of azimilide compared with placebo in prolonging the time to the first symptomatic arrhythmia recurrence in patients with a history of atrial fibrillation and congestive heart failure and/or ischemic heart disease) and those without these conditions. Once this phase of the study is completed, a second phase with a different study design will be conducted. The second phase is an open-label, follow-up phase. The follow-up phase of the study is designed to evaluate the long-term efficacy and safety of a daily oral dose of azimilide in patients who complete the double-blind, placebo-controlled phase of this study.

ELIGIBILITY:
Inclusion criteria:

* History of symptomatic atrial fibrillation that significantly disrupts the patient's customary daily living activities
* History of congestive heart failure and/or ischemic heart disease
* Sinus rhythm (normal heart rhythm) upon entry to the 30 day screening period for the study
* At least one episode of symptomatic atrial fibrillation during the screening period, with a spontaneous return to sinus rhythm.
* Sinus rhythm immediately prior to dosing

Exclusion criteria:

* Previously unsuccessful cardioversions within 60 days of screening period
* Failed to respond to any Class III antiarrhythmic drugs
* Qualifying arrhythmia due to acute reversible illness, acute myocardial infarction, and/or cardiac or thoracic surgery within one month prior to randomization
* Previously in an azimilide study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2000-12; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
To prolong the tachycardia-free period in patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Phillips, MD, Study Director — Procter and Gamble
Locations (103):
- United States (88):
  - Cardiovascular Assoc. PC, Birmingham, Alabama
  - The Heart Group, PC, Mobile, Alabama
  - Southern Arizona VA Health Care System, Section of Cardiology (1-111C), Tucson, Arizona
  - University Medical Center, Tucson, Arizona
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Cardiovascular Associates of Penisula, Burlingame, California
  - Capitol Interventional Cardiology, Carmichael, California
  - VA Central California Health Care System, Fresno, California
  - Valley Research, Fresno, California
  - Grass Valley Cardiology, Grass Valley, California
  - San Diego Cardiovascular Associates, La Jolla, California
  - Good Samaritan Hospital, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - Cardiology Section, West Los Angeles VA Hospital, Los Angeles, California
  - Merced Heart Associates, Merced, California
  - Sutter Gould Medical Foundation, Modesto, California
  - ARI Clinical Trials, Redondo Beach, California
  - Regional Cardiology Assoc., Sacramento, California
  - Sacramento Heart and Vascular Medical Associates, Sacramento, California
  - Cardiology Associates, San Diego, California
  - Aurora Denver Cardiology, Aurora, Colorado
  - Western Cardiology Assoc., Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The George Washington University MFA, Washington D.C., District of Columbia
  - Cardiology Consultants, Daytona Beach, Florida
  - C/O Research Office Attn: Cardiovascular Research Dept., Fort Lauderdale, Florida
  - SW Florida Heart Group/Health Park Medical Center, Fort Myers, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Watson Clinic, LLP, Lakeland, Florida
  - Khalid Hassan Sheikh 80 Fontenberry Road, Merritt Island, Florida
  - Florida Cardiology, Orlando, Florida
  - Cardiology Research Assiocates, Ormond Beach, Florida
  - VA Medical Center, Decatur, Georgia
  - Mount Sinal Hospital Medical Center, Chicago, Illinois
  - Elgin Cardiology Associates, Elgin, Illinois
  - Illinois Heart & Lung Research Center, SC, Normal, Illinois
  - The Center for Advanced Cardiology, Park Ridge, Illinois
  - Heart Center Medical Group, Fort Wayne, Indiana
  - The Care Group, Indianapolis, Indiana
  - Professional Research Network of Kansas, Wichita, Kansas
  - University of Louisville-Cardiology, Louisville, Kentucky
  - Louisville Cardiology Medical Group, P.S.C, Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Richard Gilmore, MD 501 S Ryan Street, Lake Charles, Louisiana
  - Cardiovascular of the South, Morgan City, Louisiana
  - Cardiovascular Institute of the South, New Iberia, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Cardiovascular Institute of the South, Thibodaux, Louisiana
  - Maine Medical Center, Portland, Maine
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusett, Worcester, Massachusetts
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Nisus Research, Petoskey, Michigan
  - Riverside Osteopathic Hospital, Trenton, Michigan
  - Regional Heart Center, Duluth, Minnesota
  - Fairview Range Regional Health Services, Hibbing, Minnesota
  - VA Medical Center Therapeutic Section, Minneapolis, Minnesota
  - St. Patrick Hosp/Western Mt. Clinic Cardiology, Missoula, Montana
  - Internal Medical Associates, Grand Island, Nebraska
  - William Olney, MD 21 Whitehall Rd, Suite 200, Rochester, New Hampshire
  - Cardiology & Int. Medicine, Williamsville, New York
  - Duke Medical Center, Durham, North Carolina
  - Altru Health System Research Center, Grand Forks, North Dakota
  - Lindner Clinical Trial Ctr., Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - MidWest Cardiology Research Foundation, Columbus, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Hillsboro Cardiology, Hillsboro, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Heart Care Group PC, Allentown, Pennsylvania
  - Tri-State Medical Group Cardiology, Beaver, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Pavillion, Jenkintown, Pennsylvania
  - UPHS/Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Cardiovascular and Critical Care Associates, P.C., Pittsburgh, Pennsylvania
  - Charleston Cardiology, Charleston, South Carolina
  - Stern Cardiovascular Center Research Department, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Heart and Vascular Inst. of Texas, PA, San Antonio, Texas
  - MedSource, Inc, Chesapeake, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
  - Daniel Gottlieb, MD 16259 Sylvester Road SW, Suite 401, Seattle, Washington
  - Beloit Clinic, SC, Beloit, Wisconsin
  - Dean/Riverview Clinic, Janesville, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (15):
  - Heart Health Institute, Calgary, Alberta
  - Heart Health Research Center, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Cardiology Research St. Paul's Hospital, Vancouver, British Columbia
  - Neureka Research Corporation, Greater Sudbury, Ontario
  - Hamilton Health Science Corp., Hamilton, Ontario
  - Cardiac Investigation Unit, London, Ontario
  - Niagara Health System Greater Niagara General Hospital, Niagara Falls, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Recharche Cardiologie, Montreal, Quebec
  - Chum Hotel Dieu, Montreal, Quebec
  - Hospital Sacre-Soeur de Montreal, Montreal, Quebec
  - Quebec Heart Institute, Sainte-Foy, Quebec